CLINICAL TRIAL: NCT02970058
Title: Platelet-rich Plasma Use as Prophylactic of Low Back Pain Post-spinal Following Gynecological Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman A. Ismail, Lecturer of anesthesia, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 01003060392
Record Dates: First submitted 2016-11-17; First posted 2016-11-21 (Estimated); Last update posted 2020-03-16 (Actual); Status verified 2019-03

CONDITIONS: Platelet-rich Plasma in Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet-rich Plasma (Active Comparator): 30 patients will receive platelet-rich plasma post-spinal anesthesia
  Interventions: Other: Platelet-rich Plasma
- Control (Placebo Comparator): 30 patients will receive sterile saline post-spinal anesthesia
  Interventions: Other: Control

INTERVENTIONS:
Other: Platelet-rich Plasma — The active group will receive Platelet-rich Plasma following spinal injection
  Arms: Platelet-rich Plasma
Other: Control — The control group will receive saline as a placebo
  Arms: Control

SUMMARY:
Platelet-rich Plasma Use as Prophylactic of Post-operative Low Back Pain Following gynecological surgery.

ELIGIBILITY:
Inclusion Criteria:

* Elective gynecological surgery.

Exclusion Criteria:

* Spinal Pathology

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-03-07 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07-15 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt